CLINICAL TRIAL: NCT01103999
Title: Prospective Evaluation of Spleen Injury Treatments in Languedoc Roussilon, France
Brief Title: Prospective Evaluation of Spleen Injury Treatments in Languedoc Roussillon
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2009/MCL-01; 2009-A00969-48 (Other: Afssaps, RCB number)
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Trauma
Keywords: spleen
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Descriptive, prospective, multicenter evaluation of spleen injury treatment in the Languedoc Roussilon region according to trauma severity, morbi-mortality and length of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for abdominal trauma
* diagnosis of splenic contusion confirmed by scanner or during surgery for hemodynamically unstable cases
* patient has signed a consent form
* patient is a beneficiary of or affiliated with a social security program

Exclusion Criteria:

* Refuses to participate
* Pregnant or breastfeeding
* Patient under guardianship

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population includes patients hospitalized for trauma to the spleen.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
Number of deceased participants | 1 year
  Mortality

SECONDARY OUTCOMES:
Number of participants with certain morbidities | 3 months of follow up
  The occurrence of pulmonary, thrombo-embolic, hemorrhagic, pancreatic, splenic and infectious morbidities are recorded.
Days in hospital | 1 year of follow up
Direct costs (euros per patient) | 1 year of follow up
  Costs are calculated as a function of hospitalisation, surgical procedures, interventional radiology.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine Le Moine, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (12):
- France (12):
  - Centre Hospitalier d'Alès, Alès
  - CH d'Avignon - Centre Hospitalier Henri Duffaut, Avignon
  - Centre Hospitalier Général Louis Pasteur, Bagnols-sur-Cèze
  - Centre Hospitalier Général, Béziers
  - Centre Hospitalier Antoine Gayraud, Carcassonne
  - APHM - Hôpital Nord, Marseille
  - Centre Hospitalier de Mende, Mende
  - Hôpital Saint Eloi, Montpellier
  - Centre Hospitalier de Narbonne, Narbonne
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Centre Hospitalier Saint Jean, Perpignan
  - Centre Hospitalier du bassin de Thau, Sète

REFERENCES:
- [Result] Chastang L, Bege T, Prudhomme M, Simonnet AC, Herrero A, Guillon F, Bono D, Nini E, Buisson T, Carbonnel G, Passebois L, Vacher C, Le Moine MC. Is non-operative management of severe blunt splenic injury safer than embolization or surgery? Results from a French prospective multicenter study. J Visc Surg. 2015 Apr;152(2):85-91. doi: 10.1016/j.jviscsurg.2015.01.003. Epub 2015 Feb 3. PMID 25662597